CLINICAL TRIAL: NCT07328724
Title: Critical Illness Among Recipients of Hematopoietic Cell Transplantation (CARE-HCT): a Prospective, Multicenter Observational Study in China
Brief Title: Critical Illness After Hematopoietic Cell Transplantation
Acronym: CARE-HCT
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Hematology Hospital of Chinese Academy of Medical Sciences (Hematology Research Center of Chinese Academy of Medical Sciences) (Unknown); Xinqiao hospital of the third military medical university (Unknown); First Affiliated Hospital of Zhejiang University (Other); First Affiliated Hospital of Harbin Medical University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, MD, Peking University People's Hospital
Other Study IDs: 2025-z259
Record Dates: First submitted 2025-12-27; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Critical Illness; Ventilated Patients; Hematopoetic Stem Cell Transplantation; Transplant Complication
Keywords: hematopoietic cell transplantation; critical illness; management; prognosis; transplant complication
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients after hematopoietic cell transplantation: Patients who are admitted to the intensive care unit after undergoing hematopoietic cell transplantation

SUMMARY:
This is a prospective, multicenter observational trial for patients who develop critical illness after hematopoietic cell transplantation. Patients who are admitted to the intensive care unit after undergoing hematopoietic cell transplantation at the participating medical centers will be enrolled in this study. The clinical characteristics, laboratory profiles, managements, and clinical outcomes will be prospectively collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent hematopoietic cell transplantation at any of the participating medical centers.
* Patients who are admitted to ICU for the management of critical illness following hematopoietic cell transplantation.

Exclusion Criteria:

* Admitted to ICU for a reason other than critical illness (e.g., routine postoperative monitoring) and discharged within 2 days of ICU admission.
* Unavailable in-ICU clinical outcomes or absent key baseline characteristics.
* Any other conditions that, in the opinion of the investigator, can interfere with the interpretation of data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are admitted to ICU after undergoing hematopoietic cell transplantation at any of the participating medical centers.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2036-06-30 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Before ICU discharge; within 6 months after ICU discharge; and within 1 year after ICU discharge.
  Overall survival after admission to the intensive care unit.

SECONDARY OUTCOMES:
Non-relapse mortality | Before ICU discharge; within 6 months after ICU discharge; and within 1 year after ICU discharge.
  Non-relapse mortality after ICU admission.
Relapse | At ICU admission and within 1 year of ICU discharge.
  Disease relapse or progression at or after ICU admission.
Transplant complication | At ICU admission and within 1 year of ICU discharge.
  Hematopoietic-cell-transplantation-associated complications at or after ICU admission.
Organ failure | At ICU admission and within 1 year of ICU discharge.
  Organ failure occurring at or after ICU admission.
Organ support therapy | At ICU admission and within 1 year after ICU discharge.
  The use of organ support therapy at or after ICU admission.
Long-term survival data | Up to 5 years after ICU discharge.
  Overall survival, non-relapse mortality, and transplant-related mortality during long-term follow-up after ICU discharge.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Peking University People's Hospital, Beijing
  - Xinqiao hospital of the third military medical university, Chongqing
  - First Affiliated Hospital of Zhejiang University, Hangzhou
  - First Affiliated Hospital of Harbin Medical University, Harbin
  - Hematology Hospital of Chinese Academy of Medical Sciences, Tianjin
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan

IPD SHARING:
Plan to Share IPD: Undecided